CLINICAL TRIAL: NCT00697164
Title: Randomized Trial of Erythropoietin to Prevent Death From Cerebral Impairment During Severe Malaria
Brief Title: Randomized Trial of Erythropoietin During Cerebral Malaria
Acronym: EPOMAL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Claude Bernard University (Other)
Responsible Party: PICOT/MD PhD, Claude Bernard University, Malaria Research Unit
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2516114389
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Cerebral Malaria
Keywords: Malaria; Treatment; Adjunctive; Erythropoietin; Survival
MeSH Terms: conditions — Malaria, Cerebral; Malaria | interventions — Erythropoietin; epoetin beta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Patients in group I received intravenous quinine followed by oral ACT for a total period of 6 days.
  Interventions: Drug: Placebo
- 2 (Experimental): Patients in group II received antimalarial drug as in group I and in addition 1500U/kg/day of rHUEPO for the initial 3 days.
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Placebo — Saline Admission, day 1, day 2 3 days
  Arms: 1
Drug: Erythropoietin — Erythropoietin, 1500 U/kg/day Admission, day 1, day 2 3 days
  Other Names: Neorecormon
  Arms: 2

SUMMARY:
Malaria remains one of the most common life-threatening illnesses in the tropics with a dramatic toll of more than one million deaths each year. A majority of malaria cases are non-complicated and only few evolve towards severe malaria resulting from the combination of parasite-specific virulence factors and host inflammatory responses. Cerebral malaria (CM) kills more than 1 million African children each year. CM carries a fatality rate of about 20% in adults, higher in children, despite timely and adequate chemotherapy. Moreover, the more rapid clearance of parasitaemia with new antimalarial drugs is not associated with improved survival, suggesting the potential interest for adjunctive therapies in the early phase of the disease.

Cerebral malaria leading to seizure and coma is associated with severe intracranial hypertension caused by brain-swelling. Recent imaging and post-mortem findings in adult cerebral malaria have confirmed the presence of diffuse cerebral oedema with thalamic and cerebellar white matter hypoattenuation, diffuse petechial hemorrhages and symmetric ischemic changes involving the thalamus and the cerebellum. However, the nature of the pathogenetic processes leading to cerebral malaria is incompletely understood but mechanisms linking cytokines with endothelial cells activation in the cerebral microvasculature have been recently stressed. The effect of new neuroprotective therapies has not yet been investigated, although the manifestations of cerebral malaria partly share features with neurological stroke or acute non-specific neurological disorders. The hormone erythropoietin (EPO) is probably one of the more enthusiastic drugs in this area.

EPO is as a member of type I cytokine superfamily with multiple functions, including a prominent role for erythropoiesis and neuroprotection. Systematically administered EPO crosses the blood brain barrier via the abundant expression of EPO receptors at brain capillaries, and acts as an anti-apoptotic and cytoprotective cytokine. Moreover, EPO prevents inflammation by inhibiting pro-inflammatory cytokines including TNFα, preserves endothelial cells integrity and prevents blood-brain barrier permeability. We propose a randomized clinical trial to investigate the safety and efficacy of EPO in patients presenting cerebral malaria and hospitalized at Gabriel Toure hospital, Bamako, Mali, to reduce the incidence of premature death in hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 months and 14 years old
* Severe cerebral malaria due to Plasmodium falciparum
* Coma (Blantyre score <3)
* Enlightened assessment

Exclusion Criteria:

* Any case of participation refusal
* Presence of another obvious affection being able to explain the state of the patient
* Negative malaria test (thick smear / thin smear)
* Severe anaemia

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-12 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Survival | day 5 post-inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Stephane PICOT, MD PhD, Principal Investigator — Claude Bernard University, Malaria Research Unit
Locations (1):
- Gabriel Toure Hospital, Bamako, Mali

REFERENCES:
- [Background] Bienvenu AL, Ferrandiz J, Kaiser K, Latour C, Picot S. Artesunate-erythropoietin combination for murine cerebral malaria treatment. Acta Trop. 2008 May;106(2):104-8. doi: 10.1016/j.actatropica.2008.02.001. Epub 2008 Feb 15. PMID 18359468
- [Derived] Picot S, Bienvenu AL, Konate S, Sissoko S, Barry A, Diarra E, Bamba K, Djimde A, Doumbo OK. Safety of epoietin beta-quinine drug combination in children with cerebral malaria in Mali. Malar J. 2009 Jul 24;8:169. doi: 10.1186/1475-2875-8-169. PMID 19630971